CLINICAL TRIAL: NCT03809286
Title: The Effect of rTMS to the Prefrontal Cortex in Alcohol Use Disorder
Acronym: MAGNA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Wai, Addiction Psychiatry Clinical & Research Fellow, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7691; 1K23AA028295 (NIH); 5R21AA026049 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: rTMS; alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: active vs. sham stimulation
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Stimulation (Experimental): Participants will be receiving active rTMS.
  Interventions: Device: active rTMS; Behavioral: Inpatient admission
- Sham Stimulation (Sham Comparator): Participants will be receiving sham stimulation with a smaller coil housed within the rTMS device.
  Interventions: Behavioral: Inpatient admission; Device: sham rTMS

INTERVENTIONS:
Device: active rTMS — rTMS delivers magnetic stimulation to the brain by using an electromagnet to generate a current that can penetrate the scalp and skull.
  Arms: Active Stimulation
Behavioral: Inpatient admission — All subjects will be admitted to the hospital for a brief detoxification period followed by 3 weeks of abstinence.
Device: sham rTMS — The sham coil setting is designed to mimic the auditory artifact and the scalp sensations evoked by the real coil, and to produce activation of facial muscles similar to the effect of a real H coil, without stimulating the brain itself.
  Arms: Sham Stimulation

SUMMARY:
The goal of this study is to investigate a treatment approach for alcohol use disorder (AUD) using a novel form of brain stimulation called deep repetitive transcranial magnetic stimulation (rTMS). The investigators will be targeting frontal regions of the brain that are important for memory and decision making. These brain regions have been shown to be impaired in patients with AUD. Previous studies have mostly used rTMS to a different frontal brain region that is not as deep. These studies have shown that rTMS can reduce craving for alcohol, but there is a lack of research showing that rTMS impacts alcohol consumption.

DETAILED DESCRIPTION:
This study aims to examine the effect of rTMS on alcohol drinking behavior in an observed laboratory setting. Participants with AUD will be recruited and admitted to the inpatient unit for the whole study. After a brief detoxification period, they will receive 3 weeks of rTMS while in the research unit. Before and after the 3 weeks of stimulation, participants will participate in a decision-making experiment where they can choose to have an alcoholic drink or the equivalent amount of money that the drink would cost (alcohol self-administration sessions). The investigators will examine their response to alcohol, as well as their performance on tasks that relate to impulsivity and memory. Participants will also undergo an MRI scan (with spectroscopy) before and after the stimulation period to look at changes in the medial prefrontal cortex of the brain. Participants will then meet with a study physician for 6 weeks after the study for assessments of alcohol use and medical management sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Current moderate to severe alcohol use disorder, per DSM-5
2. Use of alcohol which parallels or exceeds the amount alcohol that will be administered in this study (1 drinking episode per week raising BAL to 0.03 g/dl - approximately 2 drinks within an hour).
3. Age 22-55
4. Able to give informed consent, and comply with study procedures
5. Medically healthy, with the absence of current or past medical or neurological illnesses (including glaucoma, increased intracranial pressure, liver disease, cardiac disease, or seizure disorders)

Exclusion Criteria:

1. Has a contraindication to MRI, such as magnetically reactive implants, which includes metal in head except in mouth (cochlear implant, implanted brain stimulators, aneurysm clips), cardiac pacemakers, implanted neurostimulators and medication pumps, and intracardiac lines.
2. Substance use disorder with substances other than alcohol or nicotine. The current use of sedative-hypnotics or opiates will be exclusionary
3. Meets DSM-5 criteria for other psychiatric illness, such as major depression, that would interfere with participation.
4. History of seizures of any type
5. A family history of epilepsy
6. Taking psychotropic medication that would affect resting motor threshold (such as anticonvulsants) or increase risk of seizure (especially tricyclic antidepressants of neuroleptics)
7. Current suicide risk or a history of suicide attempt within the past 2 years
8. Have unstable physical disorders, including those that are previously undiagnosed, untreated, inadequately treated, or active to an extent which might make participation hazardous. For example, hypertension (a resting blood pressure > 140/90), heart failure, a recent history of myocardial infarction, previous stroke, brain lesions, any history of seizures under any circumstances or low hemoglobin.
9. Currently pregnant
10. History of severe alcohol withdrawal requiring medical care, such as withdrawal seizures, delirium tremens, withdrawal necessitating medical detoxification.
11. A desire to pursue standard treatment for AUD, such as a rehabilitation program or FDA approved medications for AUD

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the choice to self-administer alcohol in the laboratory as assessed by counting the number of drinks consumed in the 2-hour laboratory session. | 4 weeks
  Participants will participate in alcohol self-administration sessions in which they are presented with the choice of alcohol or money. The investigators will study the change in choices to choose alcohol during these sessions. There will be one session prior to rTMS and one after 3 weeks of rTMS.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0. | 10 weeks
  Adverse events will be assessed in recorded in accordance with CTCAE v4.0.

SECONDARY OUTCOMES:
Change in craving for alcohol measured using the Alcohol Urge Questionnaire (AUQ). | 4 weeks
  This AUQ (Bohn et al. 1995) is an 8-item self report questionnaire where participants rate a seven-point Likert scale with responses ranging from "strongly disagree" to "strongly agree", and a total score is derived from the sum of these items following reverse scoring of two items. A lower score is a better outcome which represents less desire to drink. Scores range from 8-56.
Change in GABA in the mPFC and ACC as measured with magnetic resonance spectroscopy (MRS). | 4 weeks
  MRS is performed by using an MRI machine to study metabolites and neurotransmitters in the brain.
Change in abstinence from alcohol following discharge assessed with the Time Line Follow Back Interview. | 10 weeks
Changes in cognitive control as measured by using the Frontal Assessment Battery (FAB). | 4 weeks
  The FAB is a brief tool that discriminates between frontal-temporal type cognitive issues from from Alzheimer's type memory issues. Higher scores are better and scores range from 0-18.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wai, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No